CLINICAL TRIAL: NCT05634850
Title: A Pilot Study: A Prospective, Longitudinal, Observational Study, Evaluating the Usability of the Product Kinder System Trial, Home Based Hormone for In-Vitro Fertilization (IVF) Monitoring System.
Brief Title: Evaluating the Usability of the Product Kinder System Trial, Home Based Hormone for In-Vitro Fertilization (IVF) Monitoring System.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Planet Innovation (Industry)
Responsible Party: Sponsor
Other Study IDs: 470_1036
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Kinder — Participants will test at their urine with at home with in the device. Results are sent via an app back to the clinic for reporting.

SUMMARY:
In-vitro fertilisation (IVF) treatment involves women undergoing hormone stimulation (drug dosing) to produce more oocytes (eggs) to increase their chances of fertilisation. The information that IVF clinicians currently collect on a woman's hormonal response to IVF drug dosing comes from in-clinic blood testing. This requires patients to make a visit to the IVF clinic every few days to have the blood samples taken. The blood is then analysed in a laboratory for the hormone levels and the results are then sent back to the clinic. This monitoring process of frequent onsite visits and blood draws can often be quite inconvenient and disruptive for patients.

This observational study will assess a non-invasive in vitro diagnostic (IVD) device for measuring the common fertility hormones in urine. The test system is for use by both healthcare professionals in a clinical setting and nonprofessionals in a home care setting under the guidance of a health care professional. This study will provide pilot data on the usability of the IVD device from the intended end users as well as the correlation of urinary metabolite levels as measured by the IVD device and the serum concentration as measured by blood analysers.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing controlled ovarian stimulation treatment
* 30 to 40 years old (inclusive)
* Willingness to comply with study procedures for collection and testing of urine

Exclusion Criteria:

* Illiterate in English
* No access to smart phone that is compatible with App and/or is not connected to the internet
* Patients who are diabetic (Type I and Type II), have insulin resistance or a renal/liver disorder
* Patients who have taken oral contraceptives up to 4 days before the first stimulation day of the cycle

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only as device test female fertility hormones
Study Population: Women aged 30-40 years older undergoing a controlled ovarian stimulation cycle as part of assisted reproductive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-06-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the usability of Kinder by patients undergoing controlled ovarian stimulation cycle | A single controlled ovarian stimulation cycle, typically up to 20 days
  Patients will perform tests with the Kinder system and complete a usability questionnaire on their experience.
Correlation of fertility hormone serum and urinary metabolites | A single controlled ovarian stimulation cycle, typically up to 20 days
  Correlation of E2, P4 and LH and their urinary metabolites (E1-3G, PdG and LH)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No